CLINICAL TRIAL: NCT02683213
Title: Establishing the Effect(s) and Safety of Fluoxetine Initiated in the Acute Phase of Stroke
Brief Title: Efficacy of Fluoxetine - a Trial in Stroke
Acronym: EFFECTS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: The Swedish Research Council (Other Government); Swedish Heart Lung Foundation (Other); Stroke-Riksförbundet (Unknown); Konung Gustaf V:s och Drottning Victorias Frimurarestiftelse (Unknown); Hjärnfonden (The Swedish Brain foundation) (Unknown); The Swedish Medical Association (Other)
Responsible Party: Principal Investigator, Erik Lundström, MD, PhD, MD, PhD, Senior Consultant in Neurology, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFFECTS2012; 2011-006130-16 (EudraCT Number)
Record Dates: First submitted 2016-02-02; First posted 2016-02-17 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Stroke
Keywords: fluoxetine; outcome; depression; plasticity
MeSH Terms: conditions — Stroke; Depression | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fluoxetine (Active Comparator): One capsule Fluoxetine 20mg once daily for 6 months.
  Interventions: Drug: Fluoxetine
- Placebo (Placebo Comparator): One matching capsule placebo once daily for 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluoxetine — Fluoxetine 20mg once daily for 6 months.
  Arms: Fluoxetine
Drug: Placebo — Matching placebo.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate whether routine administration of fluoxetine 20mg once daily in the 6 months initiated during the acute stroke improves the patient's functional outcome.

EFFECTS is an investigator lead Sweden-based, multicenter, parallel group, double blind placebo controlled trial with broad entry criteria and follow up at 6 and 12 months.

EFFECTS managed to recruit its anticipated numbers of 1,500 participants between 20th October 2014 and 28th June 2019. Data will be unblinded when the 6-months follow-up is completed, and the primary outcome is due to report on May 2020.

DETAILED DESCRIPTION:
Stroke is a serious, life-threatening medical condition that happens when the blood supply to a part of the brain is cut off, usually due to a blood clot (ischemic) or hemorrhage. Symptoms vary according to how much of the brain is affected and where in the brain the stroke occurs but includes paralysis, muscle weakness and speech problems.

A stroke can also have an impact on the sufferers emotions and can lead to anxiety, depression and personality changes. Fluoxetine (otherwise known as Prozac) has been used for many years to treat depression. However, there is evidence to suggest that it may also have other effects of the brain and enhance brain plasticity (the reorganisation of neural pathways in the brain) in a number of different ways.

One small study, for example, has shown that, if taken soon after a stroke, fluoxetine might improve the recovery of arm strength and lead to greater restoration of movement of the limbs.

Adult participants (at least 18 years old) who have had a stroke (either ischemic or hemorrhagic) within the last 2-15 days and still have some residual problems caused by the stroke e.g. weakness, or problems with their speech (speech impairment).

Participants are randomly allocated into one of two groups. Those in group 1 are given fluoxetine capsules for 6 months. Those in group 2 are given a placebo capsules for 6 months.

The participants are contacted after one week of starting their treatment, and then again after one month, to check on their well-being and that they are still taking their allocated caplets. Each participant is asked about any side effects and how much training they have had with e.g. a physiotherapist, occupational- or speech-therapist.

The research team contacts each participant at 3 months to check whether they are still taking the capsules, ask about bad side effects, and about how they are feeling (mood). If all is well, the participant is given enough medication to cover the rest of the study period.

The participant is asked to stop the study medication after 6 months and repeat assessments that they did before they started the study at the local hospital. They are also asked to fill in questionnaires together with their next of kin or carer. These questionnaires are sent to the trial main centre. If needed, they can also be filled in with the help of a trial nurse over the telephone.

The participants are contacted again one month after they have stopped the medication to see how they have progressed.

At 12 months after recruitment, participants are asked to complete the same questionnaires again about how well they have recovered from their stroke and what problems they now have after the stroke e.g. weakness in limbs, memory problems, problems with speech, low mood. These questionnaires can again be completed on paper or by telephone. The researchers then collect data on long-term recovery through national statistics.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent can only be obtained from a patient who according to the trial investigator is mentally capable of decision-making and who, after having received information and got answers to their questions, wants to participate in the trial.
* Brain imaging is compatible with intra cerebral hemorrhage or ischemic stroke.
* Randomization can be performed between 2 and 15 days after stroke onset and by the research group at the patient's local/emergency hospital.
* Persisting focal neurological deficit is present at the time of randomization severe enough to warrant treatment from the physicians and the patient's and relative's perspective.

Exclusion Criteria:

* Subarachnoidal hemorrhage except where secondary to a primary intracerebral hemorrhage.
* Unlikely to be available for follow up for the next 12 months e.g. no fixed home address.
* Unable to speak Swedish and no close family member available to help with follow up forms.
* Other life threatening illness (e.g. advanced cancer) that will make 12-month survival unlikely.
* History of epileptic seizures.
* History of allergy or contraindications to fluoxetine including: Hepatic impairment (S-ASAT/ALAT > 3 upper normal limit) and renal impairment (S-Creatinine levels > 180 micromol/L).
* Pregnant or breastfeeding, women of childbearing age not taking contraception. Minimum contraception is an oral contraceptive. An HCG-test is to be made prior randomization and after the end of trial medication.
* Previous drug overdose or attempted suicide.
* Already enrolled into a CTIMP.
* Current or recent (within the last month) depression requiring treatment with an SSRI antidepressant.

Current use of medications which have serious interactions with fluoxetine Use of any mono-amino-oxidase inhibitor (MAOI) during the last 5 weeks. Co-administration of Fluoxetine and a mono-amino-oxidase inhibitor (MAOI) may result in life threatening interactions. Therefore, patients on MAOI are ineligible for the EFFECTS trial. Also, any patient in need of treatment with a MAOI must stop their trial treatment for at least 5 weeks before commencing the MAOI, or to be treated as in-patients by a psychiatrist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2014-10-20 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Functional status, measured with the modified Rankin scale. | 6 months
  The simple modified Rankin scale questionnaire delivered by postal questionnaire, or via interview over the telephone or face to face to determine the modified Rankin scale.

SECONDARY OUTCOMES:
Survival | This will be determined by following patients up for 12 months.
  Survival will be analysed with the Cox proportional hazards model adjusting for the factors included in the minimisation algorithm
Functional status, measured with the modified Rankin scale. | 12 months
  The simple modified Rankin scale questionnaire delivered by postal questionnaire, or via interview over the telephone or face to face to determine the modified Rankin scale. The study will also investigate if the benefits of Fluoxetine remains at 12 months.
Health status measured with the Stroke Impact Scale | At 6 and 12 months
  Health status will be measured with the Stroke Impact Scale
Arm, hand, leg and foot strength assessed with the Stroke Impact Scale | At 6 and 12 months
  The Stroke Impact Scale will provide an overall assessment of patient outcome as well as allowing us to assess the effect of treatment on specific outcomes of importance to the patients. The Stroke Impact Scale was developed with input from both patients and caregivers and includes 8 domains (strength, hand function, ADL/IADL, mobility, communication, emotion, memory and thinking, participation) from across the full impairment-participation continuum.
  The 8 domains in the Stroke Impact Scale will be used for secondary outcome measures 5 to 13.
Hand function assessed with the Stroke Impact Scale | At 6 and 12 months
  The Stroke Impact Scale will provide an overall assessment of patient outcome as well as allowing us to assess the effect of treatment on specific outcomes of importance to the patients. The Stroke Impact Scale was developed with input from both patients and caregivers and includes 8 domains (strength, hand function, ADL/IADL, mobility, communication, emotion, memory and thinking, participation) from across the full impairment-participation continuum.
Mobility assessed with the Stroke Impact Scale | At 6 and 12 months
  The Stroke Impact Scale will provide an overall assessment of patient outcome as well as allowing us to assess the effect of treatment on specific outcomes of importance to the patients. The Stroke Impact Scale was developed with input from both patients and caregivers and includes 8 domains (strength, hand function, ADL/IADL, mobility, communication, emotion, memory and thinking, participation) from across the full impairment-participation continuum.
Communication and understanding assessed with the Stroke Impact Scale | At 6 and 12 months
  The Stroke Impact Scale will provide an overall assessment of patient outcome as well as allowing us to assess the effect of treatment on specific outcomes of importance to the patients. The Stroke Impact Scale was developed with input from both patients and caregivers and includes 8 domains (strength, hand function, ADL/IADL, mobility, communication, emotion, memory and thinking, participation) from across the full impairment-participation continuum.
Memory and thinking assessed with the Stroke Impact Scale | At 6 and 12 months
  The Stroke Impact Scale will provide an overall assessment of patient outcome as well as allowing us to assess the effect of treatment on specific outcomes of importance to the patients. The Stroke Impact Scale was developed with input from both patients and caregivers and includes 8 domains (strength, hand function, ADL/IADL, mobility, communication, emotion, memory and thinking, participation) from across the full impairment-participation continuum.
Mood and emotions assessed with the Stroke Impact Scale | At 6 and 12 months
  The Stroke Impact Scale will provide an overall assessment of patient outcome as well as allowing us to assess the effect of treatment on specific outcomes of importance to the patients. The Stroke Impact Scale was developed with input from both patients and caregivers and includes 8 domains (strength, hand function, ADL/IADL, mobility, communication, emotion, memory and thinking, participation) from across the full impairment-participation continuum.
Daily activities assessed with the Stroke Impact Scale | At 6 and 12 months
  The Stroke Impact Scale will provide an overall assessment of patient outcome as well as allowing us to assess the effect of treatment on specific outcomes of importance to the patients. The Stroke Impact Scale was developed with input from both patients and caregivers and includes 8 domains (strength, hand function, ADL/IADL, mobility, communication, emotion, memory and thinking, participation) from across the full impairment-participation continuum.
Participation in work, leisure and social activities assessed with the Stroke Impact Scale | At 6 and 12 months
  The Stroke Impact Scale will provide an overall assessment of patient outcome as well as allowing us to assess the effect of treatment on specific outcomes of importance to the patients. The Stroke Impact Scale was developed with input from both patients and caregivers and includes 8 domains (strength, hand function, ADL/IADL, mobility, communication, emotion, memory and thinking, participation) from across the full impairment-participation continuum.
Overall rating of recovery assessed with the Stroke Impact Scale | At 6 and 12 months
  The Stroke Impact Scale will provide an overall assessment of patient outcome as well as allowing us to assess the effect of treatment on specific outcomes of importance to the patients. The Stroke Impact Scale was developed with input from both patients and caregivers and includes 8 domains (strength, hand function, ADL/IADL, mobility, communication, emotion, memory and thinking, participation) from across the full impairment-participation continuum.
Adverse events/outcomes | At 6 and 12 months
  We will specifically ask for adverse events at each follow-up time (1 week, 1 month, 3 months, 6 months and 12 months), see the outcome 16-24 below. The definition of the SAE is defined according to Good Clinical Practice. We will not register known side effects of fluoxetine, which are listed in the drug's Summary of Product Characteristics. We will not register known problems following stroke, such as pneumonia, deep vein thrombosis etc.
Depression using the Montgomery-Åsberg Depression Rating Scale (MADRS) | At 6 and 12 months
  Depression using the Montgomery-Åsberg Depression Rating Scale (MADRS) and patients scoring high have a diagnosis of depression confirmed based on the DSM-IV criteria.
Number of participants with a recurrent stroke including ischaemic and hemorrhagic strokes | At 6 and 12 months
  Number of participants with a recurrent stroke including ischaemic and hemorrhagic strokes
Number of participants with an acute coronary syndromes | At 6 and 12 months
  Number of participants with an acute coronary syndromes
Number of participants with an Epileptic seizures | At 6 and 12 months
  Number of participants with an epileptic seizures
Number of participants with an episodes of Hyponatraemia | At 6 and 12 months
  Number of participants with an episodes of hyponatraemia (<125 mmol/l)
Number of participants with an upper gastrointestinal bleeding | At 6 and 12 months
  Number of participants with an upper gastrointestinal bleeding
Number of participants with other major bleeds | At 6 and 12 months
  Number of participants with an other major bleeds includes lower GI, extracranial, intracranial but extracerebral
Number of participants with poorly controlled diabetes | At 6 and 12 months
  Number of participants with an poorly controlled diabetes including hyperglycaemia (>22 mmol/l) and hypoglycaemia
Number of participants with falls resulting in injury | At 6 and 12 months
  Number of participants with falls resulting in injury
Number of participants with new fractures | At 6 and 12 months
  Number of participants with new fractures
Fatigue measured with the vitality subscale of the Health Questionnaire | At 6 and 12 months
  Fatigue will be measured with the vitality subscale of the Health Questionnaire, equivalent to SF 36.
Cognition assessed with the Stroke Impact Scale | At 6 and 12 months
  Cognition-the Stroke Impact Scale, which incorporates an assessment of memory and thinking, is used in conjunction with with the Montreal Cognitive Assessment (MoCA)
Health-related quality of life measured with the five-level Euroqol 5D (EQ5D-5 L) | At 6 and 12 months
  Health-related quality of life measured with the five-level Euroqol 5D (EQ5D-5 L).
Cost-effectiveness and cost-utility assessed by measuring costs, survival and health related quality of life (EQ5D) | At 6 and 12 months
  Direct and indirect costs will be estimated at 3-month, 6- month and 1 year. Effects will be measured using survival and EuroQoL 5 Dimensions (EQ5D) scale, which will be estimated into a utility score. The effectiveness measure that will be used for comparison purposes, the quality adjusted life years (QALYs), will be estimated by multiplying the relevant time parameter of the comparison with the estimated utility scores.
  A societal perspective will be adapted for the analysis, and comparison of costs and effects (QALYs) will be conducted for the period of the clinical trial, as well as by adopting a lifetime perspective, where costs and QALYs will be extrapolated beyond the duration of the trial over the expected lifetime of patients. Standard statistical regressions will be used in order to calculate the expected lifetime costs and QALYs.
Physical activity | 1 week, 1 month, 3 months, and 6 months
  Physical activity will be measured using the Saltin-Grimby Physical Activity Level Scale

CONTACTS AND LOCATIONS:
Overall Officials: Erik Lundström, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Three trial investigator teams have collaboratively developed a core protocol for Fluoxetine after stroke. Minor variations have been tailored to the national setting in the UK (FOCUS), Australia and New Zealand (AFFINITY) and Sweden (EFFECTS). Each trial is run and funded independently and will report its own results. A prospectively planned individual patient data meta-analysis of all three trials will subsequently provide the most precise estimate of the overall effect of fluoxetine after stroke and establish whether any effects differ between trials and subgroups of patients.

REFERENCES:
- [Background] Mead G, Hackett ML, Lundstrom E, Murray V, Hankey GJ, Dennis M. The FOCUS, AFFINITY and EFFECTS trials studying the effect(s) of fluoxetine in patients with a recent stroke: a study protocol for three multicentre randomised controlled trials. Trials. 2015 Aug 20;16:369. doi: 10.1186/s13063-015-0864-1. PMID 26289352
- [Background] Mead GE, Hsieh CF, Lee R, Kutlubaev MA, Claxton A, Hankey GJ, Hackett ML. Selective serotonin reuptake inhibitors (SSRIs) for stroke recovery. Cochrane Database Syst Rev. 2012 Nov 14;11(11):CD009286. doi: 10.1002/14651858.CD009286.pub2. PMID 23152272
- [Background] Graham C, Lewis S, Forbes J, Mead G, Hackett ML, Hankey GJ, Gommans J, Nguyen HT, Lundstrom E, Isaksson E, Nasman P, Rudberg AS, Dennis M. The FOCUS, AFFINITY and EFFECTS trials studying the effect(s) of fluoxetine in patients with a recent stroke: statistical and health economic analysis plan for the trials and for the individual patient data meta-analysis. Trials. 2017 Dec 28;18(1):627. doi: 10.1186/s13063-017-2385-6. PMID 29282099
- [Background] Lundstrom E, Isaksson E, Wester P, Laska AC, Nasman P. Enhancing Recruitment Using Teleconference and Commitment Contract (ERUTECC): study protocol for a randomised, stepped-wedge cluster trial within the EFFECTS trial. Trials. 2018 Jan 8;19(1):14. doi: 10.1186/s13063-017-2367-8. PMID 29310679
- [Derived] Legg LA, Rudberg AS, Hua X, Wu S, Hackett ML, Tilney R, Lindgren L, Kutlubaev MA, Hsieh CF, Barugh AJ, Hankey GJ, Lundstrom E, Dennis M, Mead GE. Selective serotonin reuptake inhibitors (SSRIs) for stroke recovery. Cochrane Database Syst Rev. 2021 Nov 15;11(11):CD009286. doi: 10.1002/14651858.CD009286.pub4. PMID 34780067
- [Derived] Lundstrom E, Isaksson E, Greilert Norin N, Nasman P, Wester P, Martensson B, Norrving B, Wallen H, Borg J, Hankey GJ, Hackett ML, Mead GE, Dennis MS, Sunnerhagen KS. Effects of Fluoxetine on Outcomes at 12 Months After Acute Stroke: Results From EFFECTS, a Randomized Controlled Trial. Stroke. 2021 Oct;52(10):3082-3087. doi: 10.1161/STROKEAHA.121.034705. Epub 2021 Aug 31. PMID 34465201
- [Derived] Mead GE, Graham C, Billot L, Nasman P, Lundstrom E, Lewis S, Hankey GJ, Hackett ML, Forbes J, Dennis M; FOCUS, AFFINITY and EFFECTS trialists. Update to the FOCUS, AFFINITY and EFFECTS trials studying the effect(s) of fluoxetine in patients with a recent stroke: statistical analysis plan for the trials and for the individual patient data meta-analysis. Trials. 2020 Nov 25;21(1):971. doi: 10.1186/s13063-020-04875-1. PMID 33239053
- [Derived] EFFECTS Trial Collaboration. Safety and efficacy of fluoxetine on functional recovery after acute stroke (EFFECTS): a randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2020 Aug;19(8):661-669. doi: 10.1016/S1474-4422(20)30219-2. PMID 32702335
- [Derived] Lundstrom E, Isaksson E, Nasman P, Wester P, Martensson B, Norrving B, Wallen H, Borg J, Dennis M, Mead G, Hankey GJ, Hackett ML, Sunnerhagen KS; EFFECTS Trial Collaboration. Update on the EFFECTS study of fluoxetine for stroke recovery: a randomised controlled trial in Sweden. Trials. 2020 Feb 28;21(1):233. doi: 10.1186/s13063-020-4124-7. PMID 32111264
- [Derived] Isaksson E, Wester P, Laska AC, Nasman P, Lundstrom E. Identifying important barriers to recruitment of patients in randomised clinical studies using a questionnaire for study personnel. Trials. 2019 Oct 30;20(1):618. doi: 10.1186/s13063-019-3737-1. PMID 31666093
- See also: The EFFECTS study home page, for investigators, layman and participants in the study. Currently only available in Swedish. — http://www.effects.se